CLINICAL TRIAL: NCT06935929
Title: A Study on the Associations Between Microribonucleic Acid Gene Polymorphisms and Crohn's Disease
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2025-01-210
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Extract whole genome DNA from peripheral blood
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CD patients: Some CD patients received sufficient UST (6 mg/kg) intravenous infusion at week 0, followed by one subcutaneous (SC) dose of 90 mg UST at 8 weeks. Maintenance therapy consisted of 90 mg subcutaneous UST every 8 or 12 weeks.
  Interventions: Biological: Ustekinumab - Standard Dosage
- normal controls: no biological agents treatment

INTERVENTIONS:
Biological: Ustekinumab - Standard Dosage — Some CD patients received sufficient UST (6 mg/kg) intravenous infusion at week 0, followed by one subcutaneous dose of 90 mg UST at week 8.Maintenance therapy consisted of 90 mg subcutaneous UST every 8 or 12 weeks.
  Groups: CD patients

SUMMARY:
From January 2020 to January 2025, Crohn's disease (CD) patients and gender- and age-matched normal controls were collected from the Department of Gastroenterology, the Second Affiliated Hospital of Wenzhou Medical University. The aim of this research is to explore the associations of microribonucleic acids (miRNAs) gene polymorphisms with the risk and clinicopathological characteristics of CD, and to analyze the effects of miRNAs gene variantions on the clinical response of ustekinumab (UST) treatment in CD patients at week 8.

DETAILED DESCRIPTION:
From January 2020 to January 2025, a total of 312 CD patients and 527 gender- and age-matched normal controls were collected from the Department of Gastroenterology, the Second Affiliated Hospital of Wenzhou Medical University.The genotypes of miRNAs were determined by multiplex polymerase chain reaction-ligase detection reaction technique. Unconditional logistic regression was employed to analyze the distribution of miRNAs gene polymorphisms between CD group and normal control group, as well as their influences on the clinicopathological characteristics of CD patients. Unconditional logistic regression model was used to explore the effect of miRNAs gene variation on the clinical response of CD patients in the treatment of UST at week 8.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed CD based on comprehensive clinical, colonoscopy, histopathological, laboratory, and radiographic examination results

Exclusion Criteria:

* rheumatoid arthritis, systemic lupus erythematosus, intestinal tuberculosis, ischemic enteritis, radiation enteritis, tumors, etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There was no statistically significant difference in the gender ratio, average age, and proportion of smokers between CD group and normal control group. All study subjects are from the Zhejiang Han population who are not related by blood.
Sampling Method: Probability Sample
Enrollment: 839 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
the genotypes of miRNAs | Baseline
  multiplex polymerase chain reaction-ligase detection reaction technique

SECONDARY OUTCOMES:
clinical response of ustekinumab treatment | week 8
  the changes of Harvey-Bradshaw index (HBI)

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No